CLINICAL TRIAL: NCT00887588
Title: A 36-week, Randomized, Double-blind, Multi-center, Parallel Group, Active Controlled Study to Evaluate the Efficacy, Safety and Tolerability of LCZ696 Compared to Valsartan in Patients With Chronic Heart Failure and Preserved Left-ventricular Ejection Fraction
Brief Title: LCZ696 Compared to Valsartan in Patients With Chronic Heart Failure and Preserved Left-ventricular Ejection Fraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCZ696B2214; 2009-010208-27
Record Dates: First submitted 2009-04-22; First posted 2009-04-24 (Estimated); Results first posted 2015-08-13 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Heart Failure
Keywords: Chronic heart failure; preserved ejection fraction; cardiovascular disease; NT-proBNP; biomarkers; Heart failure with preserved left-ventricular ejection; fraction
MeSH Terms: conditions — Cardiovascular Diseases | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LCZ696 (Experimental): During a single blind, run-in period, participants received placebo. Then at randomization (double blind treatment period), participants started with 50 mg LCZ696 for 1- 2 weeks, then uptitrated to 100 mg bid for 1 -2 weeks, and thereafter, uptitrated to 200 mg bid.
  Interventions: Drug: LCZ696; Drug: Placebo
- Valsartan (Active Comparator): During a single blind, run-in period, participants received placebo. Then at randomization (double blind treatment period), participants started with 40 mg Valsartan twice daily (bid) for 1 - 2 weeks, then were uptitrated to 80 mg bid for 1 -2 weeks, and thereafter, uptitrated to 160 mg bid.
  Interventions: Drug: Valsartan; Drug: Placebo

INTERVENTIONS:
Drug: LCZ696 — 50 mg, 100 mg and 200 mg tablets
  Arms: LCZ696
Drug: Valsartan — 40 mg, 80 mg and 160 mg tablets
  Arms: Valsartan
Drug: Placebo — matching placebo to LCZ696 and Valsartan

SUMMARY:
The study will assess the effects of 36 weeks of treatment with LCZ696 compared to valsartan on N-terminal pro-Brain Natriuretic Peptide (NT-proBNP) in patients with chronic heart failure and preserved left-ventricular ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented stable chronic heart failure (NYHA II-IV):

  * LVEF ≥ 45% (local measurement, assessed by echocardiography, MUGA, CT scan, MRI or ventricular angiography)
  * the ejection fraction must have been obtained within 6 months prior to randomization or after any MI or other event that would affect ejection fraction.
* Plasma NT-proBNP > 500 pg/ml at Visit 1.
* Patients with documented stable chronic heart failure (NYHA II-IV).
* Patients receiving ACE inhibitors (ACEi), an angiotensin receptor blockers (ARB) and/or a beta blockers must be on a stable dose of these medications stable for the 1 month period prior to Visit 1.
* Patients must be on diuretic therapy prior to Visit 1 (flexible dosing is permitted).
* Patients with a controlled systolic BP, defined as a target systolic BP less than 140 mm Hg; participants with BP up to and including 160 mm Hg are eligible for enrollment if they are on three or more medications to control BP at randomization (Visit 2).
* Patients with at least one of the following symptoms at the time of screening (Visit 1):

  * Dyspnea on exertion
  * Orthopnea
  * Paroxysmal nocturnal dyspnea
  * Peripheral edema
* Patients must have an eGFR ≥ 30 ml/min/1.73 m2 at Visit 1 (calculated by the Modification of Diet in Renal Disease formula).
* Patients with a potassium ≤5.2 mmol/l at Visit 1.

Exclusion Criteria:

* Patients with a prior LVEF reading <45%, at any time.
* Patients who require treatment with both an ACE inhibitor and an ARB.
* Isolated right heart failure due to pulmonary disease.
* Dyspnea and/or edema from non-cardiac causes, such as lung disease, anemia, or severe obesity.
* Presence of hemodynamically significant mitral and /or aortic valve disease.
* Presence of hemodynamically significant obstructive lesions of left ventricular outflow tract, including aortic stenosis.
* Presence of hypertrophic obstructive cardiomyopathy.
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis, Study Director — Novartis
Locations (71):
- United States (11):
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Grand Island, Nebraska
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Hillsboro, Oregon
  - Novartis Investigative Site, Wyomissing, Pennsylvania
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Houston, Texas
- Argentina (9):
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, Ramos Mejía, Buenos Aires
  - Novartis Investigative Site, San Martín, Buenos Aires
  - Novartis Investigative Site, Corrientes, Corrientes Province
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Santa Fe, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
- Brazil (4):
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São José do Rio Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (2):
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Göttingen, Germany
- India (9):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh, India
  - Novartis Investigative Site, Mangalore, Karnataka
  - Novartis Investigative Site, Manipal, Karnataka
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Hyderabad
- Italy (7):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Cosenza, CS
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Casorate Primo, PV
  - Novartis Investigative Site, Sarzana, SP
  - Novartis Investigative Site, San Daniele del Friuli, UD
  - Novartis Investigative Site, Somma Lombardo, VA
- Netherlands (8):
  - Novartis Investigative Site, Ede, Netherlands
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Delft
  - Novartis Investigative Site, Goes
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Heerenveen
  - Novartis Investigative Site, Heerlen
  - Novartis Investigative Site, Hengelo
- Poland (4):
  - Novartis Investigative Site, Warszawa/Anin, Poland
  - Novartis Investigative Site, Piotrkow Trybunalski
  - Novartis Investigative Site, Sieradz
  - Novartis Investigative Site, Wroclaw
- Romania (4):
  - Novartis Investigative Site, Craiova, Jud. Dolj
  - Novartis Investigative Site, Craiova, Jud.Dolj
  - Novartis Investigative Site, Baia Mare
  - Novartis Investigative Site, Piteşti
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, S.-Petersburg
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Spain (6):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Alicante, Valencia
- Venezuela (2):
  - Novartis Investigative Site, Caracas, Distrito Federal
  - Novartis Investigative Site, Maracaibo, Zulia

REFERENCES:
- [Background] Solomon SD, Zile M, Pieske B, Voors A, Shah A, Kraigher-Krainer E, Shi V, Bransford T, Takeuchi M, Gong J, Lefkowitz M, Packer M, McMurray JJ; Prospective comparison of ARNI with ARB on Management Of heart failUre with preserved ejectioN fracTion (PARAMOUNT) Investigators. The angiotensin receptor neprilysin inhibitor LCZ696 in heart failure with preserved ejection fraction: a phase 2 double-blind randomised controlled trial. Lancet. 2012 Oct 20;380(9851):1387-95. doi: 10.1016/S0140-6736(12)61227-6. Epub 2012 Aug 26. PMID 22932717
- [Derived] Myhre PL, Liu Y, Kulac IJ, Claggett BL, Prescott MF, Felker GM, Butler J, Pina IL, Rouleau JL, Zile MR, McMurray JJV, Ward JH, Solomon SD, Januzzi JL. Changes in mid-regional pro-adrenomedullin during treatment with sacubitril/valsartan. Eur J Heart Fail. 2023 Aug;25(8):1396-1405. doi: 10.1002/ejhf.2957. Epub 2023 Jul 11. PMID 37401523
- [Derived] Biering-Sorensen T, Lassen MCH, Shah A, Claggett B, Zile M, Pieske B, Pieske-Kraigher E, Voors A, Shi V, Lefkowitz M, Packer M, McMurray JJV, Solomon SD; PARAMOUNT Investigators. The Effect of Sacubitril/Valsartan on Left Ventricular Myocardial Deformation in Heart Failure with Preserved Ejection Fraction (PARAMOUNT trial). J Card Fail. 2023 Jun;29(6):968-973. doi: 10.1016/j.cardfail.2023.03.019. Epub 2023 Apr 7. PMID 37031887
- [Derived] Januzzi JL Jr, Packer M, Claggett B, Liu J, Shah AM, Zile MR, Pieske B, Voors A, Gandhi PU, Prescott MF, Shi V, Lefkowitz MP, McMurray JJV, Solomon SD. IGFBP7 (Insulin-Like Growth Factor-Binding Protein-7) and Neprilysin Inhibition in Patients With Heart Failure. Circ Heart Fail. 2018 Oct;11(10):e005133. doi: 10.1161/CIRCHEARTFAILURE.118.005133. PMID 30354399
- [Derived] Zile MR, Jhund PS, Baicu CF, Claggett BL, Pieske B, Voors AA, Prescott MF, Shi V, Lefkowitz M, McMurray JJ, Solomon SD; Prospective Comparison of ARNI With ARB on Management of Heart Failure With Preserved Ejection Fraction (PARAMOUNT) Investigators. Plasma Biomarkers Reflecting Profibrotic Processes in Heart Failure With a Preserved Ejection Fraction: Data From the Prospective Comparison of ARNI With ARB on Management of Heart Failure With Preserved Ejection Fraction Study. Circ Heart Fail. 2016 Jan;9(1):e002551. doi: 10.1161/CIRCHEARTFAILURE.115.002551. PMID 26754625
- [Derived] Andersen MB, Simonsen U, Wehland M, Pietsch J, Grimm D. LCZ696 (Valsartan/Sacubitril)--A Possible New Treatment for Hypertension and Heart Failure. Basic Clin Pharmacol Toxicol. 2016 Jan;118(1):14-22. doi: 10.1111/bcpt.12453. Epub 2015 Sep 4. PMID 26280447
- [Derived] Jhund PS, Claggett BL, Voors AA, Zile MR, Packer M, Pieske BM, Kraigher-Krainer E, Shah AM, Prescott MF, Shi V, Lefkowitz M, McMurray JJ, Solomon SD; PARAMOUNT Investigators. Elevation in high-sensitivity troponin T in heart failure and preserved ejection fraction and influence of treatment with the angiotensin receptor neprilysin inhibitor LCZ696. Circ Heart Fail. 2014 Nov;7(6):953-9. doi: 10.1161/CIRCHEARTFAILURE.114.001427. Epub 2014 Oct 2. PMID 25277997
- [Derived] Santos AB, Kraigher-Krainer E, Gupta DK, Claggett B, Zile MR, Pieske B, Voors AA, Lefkowitz M, Bransford T, Shi V, Packer M, McMurray JJ, Shah AM, Solomon SD; PARAMOUNT Investigators. Impaired left atrial function in heart failure with preserved ejection fraction. Eur J Heart Fail. 2014 Oct;16(10):1096-103. doi: 10.1002/ejhf.147. Epub 2014 Aug 19. PMID 25138249
- [Derived] Kraigher-Krainer E, Shah AM, Gupta DK, Santos A, Claggett B, Pieske B, Zile MR, Voors AA, Lefkowitz MP, Packer M, McMurray JJ, Solomon SD; PARAMOUNT Investigators. Impaired systolic function by strain imaging in heart failure with preserved ejection fraction. J Am Coll Cardiol. 2014 Feb 11;63(5):447-56. doi: 10.1016/j.jacc.2013.09.052. Epub 2013 Oct 30. PMID 24184245

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 308 participants were randomized to the core 12 week period, but 7 participants were excluded due to major Good Clinical Practice (GCP) violation. Of the 261 participants who completed the core, 252 participants entered the extension period.
Pre-assignment Details: Eight participants, who completed the core, could not continue in the extension because the 36 week protocol amendment was not yet approved by health authorities; 1 participant, who completed the core, discontinued before the extension start due to an adverse event.
Period: Core Period
Arm/Group | LCZ696 | Valsartan
Started | 149 | 152
Extension Efficacy Set | 127 | 125
Full Analysis Set | 148 | 146
Arterial Stiffness Set | 86 | 94
Completed | 130 | 131
Not Completed | 19 | 21
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Adverse Event | 9 | 11
Period: Extension Period
Arm/Group | LCZ696 | Valsartan
Started | 127 | 125
Arterial Stiffness Set | 86 | 94
Completed | 121 | 120
Not Completed | 6 | 5
Not completed — Adverse Event | 4 | 4
Not completed — Death | 0 | 1
Not completed — Protocol deviation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 | Valsartan | Total
Number analyzed (Participants) | 149 | 152 | 301
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.9 (9.38) | 71.2 (8.94) | 71.0 (9.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 85 | 170
  Male | 64 | 67 | 131

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in N-terminal Pro-brain Natriuretic Peptide (NT-proBNP)
Description: Evaluation of NT-proBNP was performed by a central laboratory. Change from baseline in NT-proBNP was presented as a ratio where the ratio was calculated as the NT-proBNP value at 12 weeks over the NT-proBNP value at baseline. A ratio < 1 indicates improvement.
Time Frame: Baseline, 12 weeks
Population: Participants from the full analysis set (FAS), who had both baseline and 12 week values, were included in the analysis. The FAS consisted of all randomized participants who had baseline and at least one post-baseline efficacy measurement during the double blind period.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio: endpoint/baseline (pg/mL)
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 134 | 132
ratio: endpoint/baseline (pg/mL) | 0.83 [0.68 to 1.01] | 1.08 [0.89 to 1.32]

2. Secondary Outcome: Change From Baseline in NT-proBNP and Brain Natriuretic Peptide (BNP)
Description: Evaluation of NT-proBNP and BNP was performed by a central laboratory. Change from baseline in NT-proBNP and in BNP was presented as a ratio where the ratio for NT-proBNP was calculated as the NT-proBNP value at 36 weeks over the NT-proBNP value at baseline, and the ratio for BNP was calculated as the BNP value at 36 weeks over the BNP value at baseline. A ratio < 1 indicates improvement.
Time Frame: baseline, 36 weeks
Population: Participants from the extension efficacy set, who had both baseline and 36 week values for each parameter, were included in the analysis for that parameter. The extension efficacy set included all randomized participants who had baseline and at least one post-baseline efficacy measurement during the extension period.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio: endpoint/baseline (pg/mL)
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 127 | 125
ratio: endpoint/baseline (pg/mL)
  NT-proBNP (n=115,116) | 0.78 [0.59 to 1.02] | 0.92 [0.70 to 1.21]
  BNP (n=116,113) | 1.14 [0.88 to 1.47] | 0.95 [0.73 to 1.23]

3. Secondary Outcome: Change From Baseline in Plasma Cyclic Guanine Monophosphate (cGMP)
Description: Evaluation of cGMP was performed by a central laboratory. Change from baseline in cGMP was presented as a ratio where the ratio was calculated as the cGMP value at 36 weeks over the cGMP value at baseline. A ratio < 1 indicates improvement.
Time Frame: baseline, 36 weeks
Population: Participants from the extension efficacy set, who had both baseline and 36 week values, were included in the analysis for that parameter. The extension efficacy set included all randomized participants who had baseline and at least one post-baseline efficacy measurement during the extension period.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio: endpoint/baseline (nmol/L)
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 56 | 54
ratio: endpoint/baseline (nmol/L) | 0.90 [0.78 to 1.03] | 0.85 [0.73 to 0.99]

4. Secondary Outcome: Change From Baseline in Echocardiography (ECHO) Parameters: Left Ventricular End (LVE) Diastolic Diameter, LVE Systolic Diameter, Septal End Diastolic Thickness, Posterior LV Wall End Diastolic Thickness, Relative Wall Thickness, Left Atrial Dimension
Description: A limited two-dimensional and Doppler ECHO examination was done to assess ECHO parameters. A negative change from baseline indicates improvement.
Time Frame: Baseline, 36 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 127 | 125
cm
  LVE diastolic diameter (n=98,107) | -0.23 (0.051) | -0.19 (0.051)
  LVE systolic diameter (n=98,107) | -0.12 (0.044) | -0.11 (0.044)
  Septal end diastolic thickness (n=98,106) | 0.01 (0.020) | 0.01 (0.020)
  Post. LV wall end diastolic thickness (n=99,107) | 0.00 (0.015) | 0.01 (0.015)
  Relative wall thickness (n=98,107) | 0.02 (0.008) | 0.02 (0.008)
  Left atrial dimension (n=99,108) | -0.21 (0.043) | -0.12 (0.042)

5. Secondary Outcome: Change From Baseline in Echocardiography Parameters: LVE Diastolic Volume, LVE Systolic Volume, Left Ventricular Stroke Volume, Left Atrial Volume
Description: as for outcome 4
Time Frame: Baseline, 36 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ml
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 127 | 125
ml
  LVE diastolic volume (n=94,111) | -12.66 (2.094) | -14.31 (2.027)
  LVE systolic volume (n=95,111) | -8.49 (1.251) | -9.64 (1.215)
  LV stroke volume (n=94,111) | -4.34 (1.448) | -4.63 (1.400)
  Left atrial volume (n=96,112) | -8.08 (2.133) | -2.38 (2.057)

6. Secondary Outcome: Change From Baseline in Echocardiography Parameters: Left Ventricular Ejection Fraction
Description: as for outcome 4
Time Frame: Baseline, 36 weeks
Population: Participants from the extension efficacy set, who had both baseline and 36 week values, were included in the analysis. The extension efficacy set included all randomized participants who had baseline and at least one post-baseline efficacy measurement during the extension period.
Measure: Least Squares Mean (Standard Error); unit: Percent ejection fraction
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 94 | 111
Percent ejection fraction | 2.62 (0.778) | 2.90 (0.755)

7. Secondary Outcome: Change From Baseline in Echocardiography Parameters: Left Ventricular Mass
Description: as for outcome 4
Time Frame: Baseline, 36 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: grams (g)
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 97 | 106
grams (g) | -11.26 (4.145) | -8.00 (4.106)

8. Secondary Outcome: Change From Baseline in Echocardiography Parameters: Left Ventricular Mass Index
Description: as for outcome 4
Time Frame: Baseline, 36 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: g/m^2
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 91 | 100
g/m^2 | -3.95 (2.249) | -1.94 (2.283)

9. Secondary Outcome: Change From Baseline in Echocardiography Parameters: Left Atrial Volume Index
Description: as for outcome 4
Time Frame: Baseline, 36 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: ml/m^2
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 90 | 106
ml/m^2 | -4.02 (1.260) | -0.88 (1.237)

10. Secondary Outcome: Change From Baseline in Echocardiography Parameters: Ewave Velocity, A Wave Velocity, e' at Septal Mitral Annulus, e' at Lateral Mitral Annulus
Description: as for outcome 4
Time Frame: Baseline, 36 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: cm/s
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 127 | 125
cm/s
  E wave velocity (n=100,112) | -0.60 (2.947) | 4.12 (2.897)
  A wave velocity (n=60,68) | -0.39 (4.199) | 0.59 (4.265)
  e' at septal mitral annulus (n=79,98) | 1.00 (0.266) | 0.98 (0.260)
  e' at lateral mitral annulus (n=84,96) | 0.71 (0.307) | 0.95 (0.296)

11. Secondary Outcome: Change From Baseline in Echocardiography Parameters: Ratio of E to A Velocity, E/e' Ratio
Description: A limited two-dimensional and Doppler ECHO examination was done to assess ECHO parameters. A ratio < 1 indicates improvement.
Time Frame: Baseline, 36 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 127 | 125
ratio
  E to A velocity (n=60,68) | 0.01 (0.080) | 0.07 (0.081)
  E/e' (n=83,95) | -1.18 (0.561) | -0.75 (0.543)

12. Secondary Outcome: Change in Echocardiography Parameters: Isovolumic Relaxation Time
Description: as for outcome 4
Time Frame: Baseline, 36 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: ms
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 35 | 42
ms | 0.01 (0.002) | 0.01 (0.002)

13. Secondary Outcome: Change From Baseline in Echocardiography Parameters: Tricuspid Regurgitation Velocity
Description: as for outcome 4
Time Frame: Baseline, 36 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: m/s
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 35 | 42
m/s | -0.05 (0.081) | 0.00 (0.079)

14. Secondary Outcome: Change From Baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score and Individual Domain Summary Scores
Description: The KCCQ is a self-administered questionnaire. It contains 23 items, covering physical function, clinical symptoms, social function, self-efficacy and knowledge, and quality of life, each with different Likert scale wording, including limitations, frequency, bother, change in condition, understanding, levels of enjoyment and satisfaction. Scores are transformed to a range of 0-100, in which higher scores reflect better health status. A positive change from baseline indicates improvement.
Time Frame: baseline, 36 weeks
Population: Participants from the extension efficacy set, who had both baseline and 36 week values for each domain, were included in the analysis for that domain. The extension efficacy set included all randomized participants who had baseline and at least one post-baseline efficacy measurement during the extension period.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 127 | 125
score on a scale
  Physical limitation (n=117,114) | 9.27 (2.528) | 9.88 (2.516)
  Symptom stability (n=118,116) | 6.43 (3.171) | 7.94 (3.167)
  Symptom frequency (n=118,116) | 10.38 (2.582) | 9.16 (2.577)
  Symptom burden (n=118,116) | 9.23 (2.528) | 9.45 (2.527)
  Total symptom score (n=118,116) | 9.83 (2.386) | 9.32 (2.384)
  Self efficacy (n=118,116) | 11.24 (2.427) | 8.77 (2.419)
  Quality of life (n=118,116) | 13.13 (2.706) | 12.50 (2.702)
  Social limitation (n=113,107) | 9.99 (2.878) | 11.04 (2.936)
  Overall summary score (n=118,116) | 11.25 (2.185) | 11.31 (2.183)

15. Secondary Outcome: Percentage of Participants With Clinical Composite Assessment of Improved, Unchanged or Worsened
Description: The clinical composite assessment is defined as follows: Improved = a) participant improved (markedly or moderately) in the global assessment of disease activity with no worsening of NYHA functional class and no major adverse cardiovascular event or b) participant improved in NYHA functional class with no worsening (markedly or moderately) in the global assessment of disease activity and no major adverse cardiovascular event. Worsened = participant worsened (markedly or moderately) in the global assessment of disease activity or in NYHA functional class or experienced a major adverse cardiovascular event. Unchanged = participant does not meet the definition for improved or worsened.
Time Frame: 36 weeks
Population: Extension efficacy set: the extension efficacy set included all randomized participants who had baseline and at least one post-baseline efficacy measurement during the extension period.
Measure: Number; unit: Percentage of participants
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 127 | 125
Percentage of participants
  Improved | 41.7 | 32.8
  Unchanged | 45.7 | 53.6
  Worsened | 12.6 | 13.6

16. Secondary Outcome: Percentage of Participants With New York Heart Association (NYHA) Class I, II, II or IV
Description: The NYHA Functional Classification classifies patients' heart failure according to the severity of their symptoms. The classification is as follows: Class I: no limitation of physical activity, ordinary physical activity does not cause undue fatigue, palpitation, or dyspnea (shortness of breath); Class II: slight limitation to physical activity, comfortable at rest, ordinary physical activity results in fatigue, palpitation or dyspnea; Class III: marked limitation of physical activity, comfortable at rest, less than ordinary activity causes fatigue, palpitation or dyspnea; Class IV: unable to carry on any physical activity without discomfort, symptoms of heart failure at rest, if any physical activity is undertaken, discomfort increases.
Time Frame: baseline, 36 weeks
Population: as for outcome 15
Measure: Number; unit: Percentage of participants
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 127 | 125
Percentage of participants
  Baseline, Class I | 0.8 | 0.8
  Baseline, Class II | 78.7 | 81.6
  Baseline, Class III | 20.5 | 17.6
  Baseline, Class IV | 0 | 0
  Week 36, Class I | 12.6 | 7.2
  Week 36, Class II | 74.0 | 78.4
  Week 36, Class III | 13.4 | 14.4
  Week 36, Class IV | 0 | 0

17. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR)
Description: eGFR was calculated from the serum creatinine concentration determined by central laboratory assessment. A positive change from baseline indicates improvement.
Time Frame: baseline, 36 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73m^2
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 126 | 123
mL/min/1.73m^2 | -3.68 (1.493) | -7.14 (1.517)

18. Secondary Outcome: Change From Baseline in Serum Creatinine
Description: Evaluation of serum creatinine was performed by central laboratory. A negative change from baseline indicates improvement.
Time Frame: baseline, 36 weeks
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: µmol/L
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 127 | 125
µmol/L | 5.82 (2.136) | 10.65 (2.183)

19. Secondary Outcome: Change From Baseline in Albumin/Creatinine Ratio
Description: Evaluation of albumin/creatinine was performed by central laboratory. A ratio < 1 indicates improvement.
Time Frame: baseline, 36 weeks
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 100 | 101
ratio | 1.19 [0.85 to 1.66] | 0.74 [0.52 to 1.06]

20. Secondary Outcome: Change From Baseline in Arterial Stiffness Parameters: Brachial Systolic Blood Pressure (SBP), Brachial Diastolic Blood Pressure (DBP), Central Augmentation Pressure, Central Pressure at T1-DP, Central SBP, Central DBP, Central Mean Pressure
Description: A vascular arterial stiffness sub-study was conducted in a subset of participants. Noninvasive arterial tonometry was assessed using the Sphygmor device. Participants had arterial stiffness, pulse wave velocity and central pressures measured. A negative change from baseline indicates improvement.
Time Frame: baseline, 36 weeks
Population: Participants from the arterial stiffness set, who had values for both baseline and week 36, were analyzed. The arterial stiffness set included randomized participants who participated in the arterial stiffness sub-study.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 86 | 94
mmHg
  Brachial SBP(n=36,44) | -1.27 (3.935) | 1.47 (3.670)
  Brachial DBP (n=36,44) | 1.68 (2.279) | 0.79 (2.165)
  Central augmentation pressure (n=36,44) | -0.21 (1.824) | -0.24 (1.705)
  Central pressure at T1-DP (n=36,44) | -1.92 (2.071) | 0.02 (1.941)
  Central SBP (n=36,44) | -0.71 (3.856) | 0.86 (3.594)
  Central DBP (n=36,44) | 1.40 (2.319) | 0.24 (2.204)
  Central mean pressure (n=36,44) | 0.84 (2.565) | -0.13 (2.436)

21. Secondary Outcome: Change From Baseline in Arterial Stiffness Parameters: Heart Rate Correct Cen Aug/Pulse Ht
Description: as for outcome 20
Time Frame: baseline, 36 weeks
Population: as for outcome 20
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 36 | 43
Percent | -0.74 (2.392) | -2.16 (2.250)

22. Secondary Outcome: Change From Baseline in Arterial Stiffness Parameters: Heart Rate
Description: as for outcome 20
Time Frame: baseline, 36 weeks
Population: as for outcome 20
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 36 | 44
bpm | -0.64 (2.026) | -1.32 (1.905)

23. Secondary Outcome: Change From Baseline in Arterial Stiffness Parameters: Pulse Wave Velocity
Description: as for outcome 20
Time Frame: baseline, 36 weeks
Population: as for outcome 20
Measure: Least Squares Mean (Standard Error); unit: cm/s
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 32 | 42
cm/s | -0.44 (0.731) | -0.74 (0.631)

24. Secondary Outcome: Change From Baseline in Sitting SBP, Sitting DBP and Sitting Pulse Pressure (PP)
Description: Sitting blood pressure and sitting pulse pressure were assessed. A negative change from baseline indicates improvement.
Time Frame: baseline, 36 weeks
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 | Valsartan
Number analyzed (Participants) | 125 | 127
mmHg
  mean SBP | -7.47 (1.909) | -2.18 (1.936)
  mean DBP | -5.28 (1.188) | -1.39 (1.204)
  Pulse pressure | -2.24 (1.482) | -1.17 (1.497)

ADVERSE EVENTS:
Arm/Group | LCZ696 | Valsartan
Serious Adverse Events (participants affected / at risk) | 22/149 | 30/152
Other Adverse Events (participants affected / at risk) | 79/149 | 92/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (N=149) | Valsartan (N=152)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 2
Angina unstable (Cardiac disorders) | 3 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 3 | 2
Cardiac failure acute (Cardiac disorders) | 1 | 3
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 2 | 0
Chest discomfort (General disorders) | 1 | 0
Device malfunction (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adrenal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Hyperuricosuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 1
Femoral arterial stenosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (N=149) | Valsartan (N=152)
Anaemia (Blood and lymphatic system disorders) | 2 | 5
Angina pectoris (Cardiac disorders) | 4 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 8
Bradycardia (Cardiac disorders) | 0 | 4
Cardiac failure (Cardiac disorders) | 3 | 4
Cardiac failure chronic (Cardiac disorders) | 1 | 4
Palpitations (Cardiac disorders) | 5 | 5
Vertigo (Ear and labyrinth disorders) | 5 | 1
Cataract (Eye disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Constipation (Gastrointestinal disorders) | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 9 | 4
Dyspepsia (Gastrointestinal disorders) | 4 | 2
Nausea (Gastrointestinal disorders) | 3 | 4
Asthenia (General disorders) | 7 | 10
Fatigue (General disorders) | 3 | 6
Non-cardiac chest pain (General disorders) | 3 | 0
Oedema peripheral (General disorders) | 4 | 9
Pyrexia (General disorders) | 4 | 0
Bronchitis (Infections and infestations) | 6 | 2
Gastroenteritis (Infections and infestations) | 4 | 1
Influenza (Infections and infestations) | 4 | 5
Nasopharyngitis (Infections and infestations) | 3 | 5
Respiratory tract infection (Infections and infestations) | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 6 | 9
Dyslipidaemia (Metabolism and nutrition disorders) | 3 | 0
Gout (Metabolism and nutrition disorders) | 0 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 10 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2
Dizziness (Nervous system disorders) | 11 | 7
Headache (Nervous system disorders) | 3 | 4
Insomnia (Psychiatric disorders) | 1 | 4
Renal impairment (Renal and urinary disorders) | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 5
Hypertension (Vascular disorders) | 3 | 6
Hypotension (Vascular disorders) | 19 | 14
Orthostatic hypotension (Vascular disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.